CLINICAL TRIAL: NCT02829788
Title: Study Comparing the Role of the Laparoscopy Surgical Staging in the Peritoneal Carcinomatosis to Laparotomic Approach
Acronym: COELIOCHIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0433
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Peritoneal Carcinomatosis
Keywords: Digestive peritoneal carcinomatosis; laparoscopy; laparotomy; peritoneal cancer index (PCI); staging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Digestive peritoneal carcinomatosis staging: All patients underwent laparoscopic followed by laparotomic surgical staging.
  Interventions: Other: Non interventional

INTERVENTIONS:
Other: Non interventional — Peroperative data collection

SUMMARY:
The peritoneum is the second most common site of recurrence in patients with colorectal cancer. Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy improve the prognosis of these patients and incorporates surgical removal of all visible disease followed by chemical destruction of microscopic disease through chemoperfusion. The most validated predictors of outcome are preoperative tumor burden measured in terms of the peritoneal carcinomatosis index (PCI) and completeness of cytoreduction (CC score). Diagnostic laparoscopy prior to resection is widely used in hepatopancreaticobiliary and colorectal cancer and has been shown to be effective in excluding unnecessary laparotomy associated with higher morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Colorectal cancer with a resected minimal synchronous peritoneal carcinomatosis, or ovarian metastases, tumour rupture in the abdominal cavity.
* Patients received six months of systemic chemotherapy (currently the Folfox-4 regimen which could be modified if the standard is modified)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospectively diagnosed patients initially treated with surgery and adjuvant chemotherapy who have a high risk of developing colorectal peritoneal carcinomatosis.
  All patients will receive the current standard adjuvant treatment: 6 months of systemic chemotherapy (currently the Folfox-4 regimen which could be modified if the standard is modified). Then a work-up is done to exclude recurrence.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal carcinomatosis staging | during laparoscopy and during laparotomy (Day 1)
  To score the Collect detailed detailed Peritoneal Cancer Index (PCI) by laparoscopy following the laparotomy procedure in order to evaluate the accuracy and adequacy of laparoscopic surgical staging comparing to laparotomic approach.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GLEHEN, Prof, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud - Service de Chirurgie Générale et Digestive - 165 chemin du grand Revoyet, PIERRE-BENITE, FRANCE, 69495
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud Service de Chirurgie Générale et Digestive - 165 chemin du grand Revoyet, Pierre-Bénite, France